CLINICAL TRIAL: NCT07001930
Title: Pharmacological Effects of Cannabidiol on Responses to Stress and Nicotine Withdrawal
Brief Title: Effects of Cannabidiol on Stress and Nicotine Withdrawal
Acronym: CREWS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB00440948; R01DA027232-09A1 (NIH)
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: CBD; Stress; Nicotine Dependence; Tobacco Smoking
Keywords: CBD; Stress; Nicotine; Tobacco Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Smoking | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled, within-subjects crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ad Lib (first) (Experimental): Participants who use tobacco cigarettes and will be randomly assigned to smoking ab lib. Each participant will receive 0, 200, 400 mg of CBD in this arm.
  Interventions: Drug: Epidiolex
- Abstinence (first) (Experimental): Participants who use tobacco cigarettes and will be randomly assigned to smoking abstinence for 24 hours before each session. Each participant will receive 0, 200, 400 mg of CBD in this arm.
  Interventions: Drug: Epidiolex

INTERVENTIONS:
Drug: Epidiolex — Oral cannabidiol

SUMMARY:
The purpose of this study is to examine the effect of doses of cannabidiol (CBD) during exposure to stress and nicotine withdrawal in nicotine users. The main objectives of the study include examining the effect CBD has on stress, tobacco dependence, tobacco withdrawal, and sex differences between these types of stress. Participants will be administered CBD and exposed to stress. Biological and subjective measures will be collected. Participants may be asked to stop use for 24 hours. Researchers will also investigate withdrawal effects between participants who have not smoked nicotine in 24 hours and those who have continued to smoke before each session.

DETAILED DESCRIPTION:
This study will use a double-blind, placebo-controlled, within-subjects crossover design to examine the effect of acute doses of CBD during exposure to acute stress and nicotine withdrawal using a relevant set of biological and subjective measures that are known to be sensitive to acute stress and to nicotine withdrawal. There will be one in-person medical screening session, 3 pre-laboratory phone sessions, and 3 in-person experimental laboratory sessions separated by at least 72 hrs. Total duration for a study completer is estimated to be 2-3 weeks. Three doses of CBD (0mg, 200mg, and 400mg) will be administered, one at each of three separate laboratory sessions that will last approximately 5 hours each and be separated by at least 72 hours. Two effective induction challenges will be implemented: one is behavioral (an established and well validated acute psychological stress induction) and one is a nicotine withdrawal challenge (24 hours abstinence from all nicotine products). Nicotine users reporting daily cigarette use (N=90) will be recruited. Nicotine users will be randomly assigned to continue nicotine use ad libitum or to abstain for 24 hours before each of three laboratory sessions. Randomization will be stratified based on participant sex and current use of other tobacco products (e.g. e-cigarettes, smokeless tobacco, pouches, cigars/cigarillos). Participants who use other nicotine-related products (e.g., e-cigarettes) will be accepted in the study if they also smoke cigarettes. Use of other nicotine products will be assessed and tracked to account for their effects on the collected measures.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy non-treatment seeking adults aged 21-70 (inclusive).
2. Use of > 5 cigarettes per day for > 2 years. (Use of other tobacco/nicotine products in addition to cigarettes will be acceptable).
3. Biological confirmation of cigarette use: have an expired carbon monoxide (CO) level > 8 ppm.
4. Alcohol Use: < 2 drinks/day on average (< 14 drinks/week).
5. Sleep schedule: No graveyard or third shift work (i.e., participants must report a normal nighttime sleep schedule).
6. For women of children bearing potential and men with female partners of child-bearing potential, must be willing to use an effective form of contraception during the study and for at least 30 days after the last study drug administration.

Exclusion Criteria:

1. Report current intention to reduce or quit cannabis or tobacco use within the next 30 days
2. Meet Diagnostic and Statistical Manual (DSM-5) criteria for a substance use disorder other than alcohol, cannabis, or nicotine
3. Test positive for illicit drugs other than cannabis
4. Positive breath alcohol test (>.01 g/210L) at study admission
5. Have a current physical or mental illness or takes a medication judged by the study team to negatively impact participant safety or scientific integrity
6. Have a resting heart rate >100, systolic blood pressure >160mmHg or <100mmHg, or diastolic blood pressure >100mmHg or <50mmHg at screening.
7. Have cold intolerance or a medical condition that might be exacerbated by exposure to cold (e.g. Reynaud's, peripheral neuropathy, trigeminal neuralgia, poorly controlled/uncontrolled hypothyroidism).
8. Are currently pregnant, planning to become pregnant in the next three months, or are currently breastfeeding
9. Have a history of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina, Raynaud's).
10. Have a history of and/or current liver disease, or elevated serum liver transaminase (AST or ALT) above 3 x Upper Limit of Normal (ULN), or elevated bilirubin above 2 x ULN at screening.
11. Are currently enrolled in another clinical trial or have received any drug as part of a research study within 30 days of study participation.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Negative Affect as assessed by the Subjective State Scale | 20 minutes, 70 minutes, 120 minutes, 170 minutes, 190 minutes, 200 minutes, 220 minutes timepoints
  Negative affect is measured using the Subjective State Scale which includes 4 items measuring negative affect. The scale has a range of 0 to 28 with higher scores indicating greater negative affect.
Positive Affect as assessed by the Subjective State Scale | 20 minutes, 70 minutes, 120 minutes, 170 minutes, 190 minutes, 200 minutes, 220 minutes timepoints
  Positive affect is measured using the Subjective State Scale which includes 5 items measuring positive affect. The scale has a range of 0 to 35 with higher scores indicating greater positive affect.
Blood Plasma Cortisol level | 20 minutes, 70 minutes, 120 minutes, 170 minutes, 190 minutes, 200 minutes, 220 minutes timepoints
  Blood plasma cortisol will be collected during laboratory stress testing sessions using a 20-gauge IV Teflon catheter inserted in a non-dominant forearm vein.
Salivary Cortisol level | 20 minutes, 70 minutes, 120 minutes, 170 minutes, 190 minutes, 200 minutes, 220 minutes timepoints
  Salivary cortisol will be collected during laboratory stress sessions using Salivette tubes and assayed using time-resolved fluorescence immunoassay.
Plasma Concentration of Endocannabinoids | 20 minutes, 70 minutes, 120 minutes, 170 minutes, 190 minutes, 200 minutes, 220 minutes timepoints
  Blood plasma endocannabinoids will be collected during laboratory stress testing sessions using a 20-gauge IV Teflon catheter inserted in a non-dominant forearm vein.
Heart Rate (beats per minutes) | 20 minutes, 70 minutes, 120 minutes, 170 minutes, 190 minutes, 200 minutes, 220 minutes timepoints
  Heart rate will be collected during laboratory stress testing sessions.
Systolic Blood Pressure (mmHg) | 20 minutes, 70 minutes, 120 minutes, 170 minutes, 190 minutes, 200 minutes, 220 minutes timepoints
  Systolic blood pressure will be collected during laboratory stress testing sessions.
Diastolic Blood Pressure (mmHg) | 20 minutes, 70 minutes, 120 minutes, 170 minutes, 190 minutes, 200 minutes, 220 minutes timepoints
  Diastolic blood pressure will be collected during laboratory stress testing sessions.

SECONDARY OUTCOMES:
Subjective Pain as assessed by the McGill Pain Questionnaire short form (MPQ) | 170 minute timepoint
  Subjective pain will be measured immediately after the cold pressor task (CPT) at each stress session using the McGill Pain Questionnaire short form, with a score range of 0 to 78, with higher values indicating more significant pain.
Nicotine urge as assessed by the Questionnaire on Smoking Urges (QSU-brief) | 20 minutes, 70 minutes, 120 minutes, 170 minutes, 190 minutes, 200 minutes, 220 minutes timepoints
  Nicotine urge will be measured using the Questionnaire on Smoking Urges (QSU-brief) includes 10 items on a likert scale from 1 to 7. Total score range is 7 to 70, higher scores more nicotine urge.
Craving for Sweet and Rich Foods as assessed by the Questionnaire on Craving for Sweet and Rich Food, | 200 minute timepoint
  Craving for sweet and rich foods will be measured using the Questionnaire on Craving for Sweet and Rich Food, which includes one question assessing craving sweet or rich foods at the current moment, with scores ranging from 1 to 7, with higher scores indicating greater craving.
Hypothetical Tobacco Demand | 200 minute timepoint
  Hypothetical tobacco demand will be measured using a cigarette purchase task after each laboratory stress session. Change in demand (amplitude and persistence) will be assessed to create an overall demand curve.
Sustained Attention to Response Task | 200 minute timepoint
  Sustained attention will be measured using the Sustained Attention to Response Task. Errors of commission and errors of omission will be assessed during the recovery period at each laboratory stress session.
Reaction time on the N-Back Cognitive test | 200 minute timepoint
  N-back task (0 back and 1 back) accuracy will be used to measure working memory during the recovery period at each laboratory stress session. Participants will be exposed to a series of numbers and will be asked to respond on a keypad when the current number matches a number presented "n" trials back.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin C. Lee, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States